CLINICAL TRIAL: NCT05191615
Title: Workplace Motivation, Job-Satisfaction, and Wellness, Among Nurses and Managers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit sufficient sample size to reach power.
Sponsor: Billings Clinic (Other)
Collaborators: University of South-Eastern Norway (Other); University of Rochester (Other)
Responsible Party: Principal Investigator, Jamie Besel, Research Scientist, Billings Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21.019
Record Dates: First submitted 2021-12-16; First posted 2022-01-13 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Motivation; Job Satisfaction; Wellness
Keywords: Nurse

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled Trial (RCT) design will be used to evaluate the effect of job-crafting, need crafting, and preventative health visits based on motivational underpinnings. As a basis for collecting data through the different time points and evaluate the intervention, the study will adopt a mixed method approach. That is, both qualitative (i.e., focus groups and interviews) and quantitative (i.e., questionnaires) methods will be applied to evaluate the interventions implemented.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The proposed study will be implemented as an intervention study at two levels within the organization, managerial and registered nurses. The intervention comprises three major phases: a pre-intervention phase, an implementation-intervention phase, and a post-intervention phase. The interventions will be provided face-to-face by trained interventionists. At baseline, all participants will complete questionnaires and get labs completed, blood pressure checked, and weight/height measured.
  Consists of two main parts. In the first part, both managers and employees will be trained in the principles of SDT and JD-R. For managers, particular attention will be paid to the provision of need support and work values. For employees, particular attention will be paid to employees' opportunities for job crafting and promoting their basic psychological need satisfaction at work.
  Interventions: Behavioral: Job crafting training
- Control Group (No Intervention): Participants randomized to the control group will complete the baseline questionnaires and lab tests at baseline and three follow-up times. Lab values will be collected using the current standard of care and American Heart Association (AHA) guidelines (2019).

INTERVENTIONS:
Behavioral: Job crafting training — Consists of two main parts. In the first part, both managers and employees will be trained in the principles of SDT and JD-R. For managers, particular attention will be paid to the provision of need support and work values. For employees, particular attention will be paid to employees' opportunities for job crafting and promoting their basic psychological need satisfaction at work.
  In the second part of the intervention, participants will have the opportunity to discuss their current health status and receive preventive health recommendations from a preventive care specialist.
  Arms: Intervention Group

SUMMARY:
The purpose of this research project is to assess the impact of a multi-level intervention designed to optimize work motivation and support physical and psychological health among employees. The intervention is based on the principles of self-determination theory; an empirically based approach to human motivation that has been applied to work and health and the job demands resources (JD-R) model; an empirically based model of occupational health.

DETAILED DESCRIPTION:
This study will provide insight into the work climate conditions that are necessary to promote healthy, productive employees and organizations. Based on the knowledge gaps identified in the literature, this will be done by examining the motivational underpinnings related to this challenge to understand the temporal processes leading workplace factors to various occupational health consequences and organizational performance.

1. Aim 1: Develop, implement, and evaluate the effectiveness of a one-and-a-half-day training for nurse managers on 1) how to provide need support 2) facilitate job crafting and 3) how to conduct values interviews to employees (i.e., staff nurses). Following the training, managers will be prepared to implement a need-supportive style during interactions with employees and conduct a values interview.
2. Aim 2: Develop, implement, and evaluate the effectiveness of an intervention for staff nurses to include 1) a one-day training on job crafting and need crafting at work with weekly boosters; 2) a values interview with their manager; and 3) a preventive health assessment and intervention.

ELIGIBILITY:
Inclusion Criteria:

* • Registered Nurse, Manager, or Clinical Supervisor employed at the hospital.

  * Employed by Billings Clinic for a minimum of 6 months.
  * Plan to be in the community for 12-18 months.
  * Proficiency in spoken and written English.

Exclusion Criteria:

* • New employee, defined as <6 months employment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in basic psychological need satisfaction at work | Baseline, 3 months, 6 months, 9 months, 12 months
  Self-Determination Theory (SDT) identifies three basic psychological needs that must be supported for humans to be optimally healthy, at work or otherwise. These needs are for autonomy (the need to feel volition and to endorse one's behavior), competence (that one can achieve desired outcomes), and relatedness (that one feels warmly and positively connected to others).
Change from Baseline in Managerial Autonomy Support | Baseline, 3 months, 6 months, 9 months, 12 months
  The Work Climate Questionnaire, Short Form (Baard et al. 2004; Schultz et al., 2015) assessed perceptions of autonomy support from the participant's most immediate supervisor over the past 4 weeks. The scale comprises six items, and responses were made on a 7- point scale from 1 (strongly disagree) to 7 (strongly agree), with higher scores indicating greater perceived managerial autonomy support. Sample items include "My supervisor tries to understand how I see things before suggesting a new way to do things" and "I feel that my supervisor provides me with choices and options." Reliability in this sample was good, α=0.94.
Change from Baseline in Organizational need support | Baseline, 3 months, 6 months, 9 months, 12 months
  6-item questionnaire that contains items related to employee experience at the organization.
Change from Baseline in Work motivation | Baseline, 3 months, 6 months, 9 months, 12 months
  Questionnaire that assesses external regulation, introjection, identified regulation, intrinsic motivation, and amotivation at work. Response scale: 1 (not at all for this reason), 2 (not really for this reason), 3 (a little for this reason), 4 (moderately for this reason), 5 (strongly for this reason), 6 (very strongly for this reason), 7 (exactly for this reason)
Change from Baseline in Job crafting | Baseline, 3 months, 6 months, 9 months, 12 months
  Questionnaire assessing how often the employee engages in the following behaviors; optimizing hindering demands, increasing structural resources, increasing social resources, increasing challenging demans, and reframing job conception.
Change in Baseline in Need crafting | Baseline, 3 months, 6 months, 9 months, 12 months
  Questionnaire assessing how often the employee engages in the following behaviors of autonomy crafting, competence crafting, and relatedness crafting. The response scale: 1 (never), 2 (rarely), 3 (sometimes), 4 (often), 5 (very often).
Change in Baseline in Work value orientations | Baseline, 3 months, 6 months, 9 months, 12 months
  Questionnaire assessing intrinsic work values and extrinsic work values. Response scale: 1 (very unimportant), 2 (slightly unimportant), 3 (neutral), 4 (slightly important) 5 (very important)
Change in Baseline in Work characteristics | Baseline, 3 months, 6 months, 9 months, 12 months
  Questionnaire that assesses characteristics of the job including skill variety, task variety, job feedback, job autonomy, social feedback, social impact, role conflict, workload, emotional demands, and cognitive demands. Response scale: 1 (strongly disagree) to 5 (strongly agree)
Change in Baseline in Work stress and burnout | Baseline, 3 months, 6 months, 9 months, 12 months
  Questionnaire assessing the amount of stress felt at work and how often burnout is experienced. Response scale: 0 (never), 1 (a few times a year or less), 2 (once a month or less), 3 (a few times a month), 4 (once a week), 5 (a few times a week), to 6 (every day)
Change in Baseline in Vigor | Baseline, 3 months, 6 months, 9 months,12 months
  Questionnaire assessing energy and vigor over the past year. Response scale: 0 (never), 1 (a few times a year or less), 2 (once a month or less), 3 (a few times a month), 4 (once a week), 5 (a few times a week), to 6 (every day)
Change in Baseline in work performance | Baseline, 3 months, 6 months, 9 months, 12 months
  Questionnaire assessing employee performance over the past year and includes task proficiency, task adaptivity, task proactivity. Response scale: 1 (very little) to 5 (a great deal).
Change in Baseline in Turnover intention | Baseline, 3 months, 6 months, 9 months, 12 months
  Questionnaire that assesses employee view of job change. Response scale: 1 (never), 2 (very rarely), 3 (rarely), 4 (sometimes), 5 (often), 6 (often), 7 (all the time).
Change in Baseline in job and life satsifaction | Baseline, 3 months, 6 months, 9 months, 12 months
  Assesses overall satisfaction with the job and life; a total of 2 questions. Response scale: 1 (strongly disagree), 2 (disagree), 3 (slightly disagree), 4 (neither agree nor disagree), 5 (slightly agree), 6 (agree), 7 (strongly agree).

SECONDARY OUTCOMES:
Change in Baseline in somatic symptom burden | Baseline, 3 months, 6 months, 9 months, 12 months
  Using a response scale of 0 (not at all) to 4 (very much), participants are asked how much they have been bothered by 8 different symptoms during the past 4 weeks.
Change in Baseline in Clinician need support | Baseline, 3 months, 6 months, 9 months, 12 months
  Participants will be asked to rate their agreement on a scale of 1-5, with 5 meaning strongly agree and 1 meaning strongly disagree.
Change in baseline Autonomous motivation for a Heart Healthy Lifestyle and Medications to Optimize My Health | Baseline, 3 months, 6 months, 9 months, 12 months
  Participants are sked to rate their agreement on a scale of 1-5 regarding their motivation toward a heart healthy lifestyle.
Change in Baseline in Perceived competence for living a heart healthy lifestyle. | Baseline, 3 months, 6 months, 9 months, 12 months
  This questionnaire asks participants to rate their agreement on a scale of 1-5 regarding their perceived competence for living and maintaining a heart healthy lifestyle.
Change in Baseline in Quality of Lide | Baseline, 3 months, 6 months, 9 months, 12 months
  Participants are asked one question each regarding their general health status, physically unhealthy days, mentally unhealthy days, and activity limitation days.
Change in Baseline in Sleep quality | Baseline, 3 months, 6 months, 9 months, 12 months
  Participants are asked if they've experienced sleep issues during the past month. A total of 2 questions are asked using the response scale 1 (never), 2 (sometimes), 3 (often, 4 (almost every night).
Change in baseline in alcohol use | Baseline, 3 months, 6 months, 9 months, 12 months
  Participants are asked about average days per week they drink alcohol and the amount.
Change in Baseline Physical Activity | Baseline, 3 months, 6 months, 9 months, 12 months
  Assess how many times a week the participant does vigorous and moderate physical activity.
Change in Baseline in fruit and vegetable intake | Baseline, 3 months, 6 months, 9 months, 12 months
  Assesses over the last month how many pieces of fruit and vegetables eaten.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie M Besel, PhD, Principal Investigator — Billings Clinic
Locations (1):
- Billings Clinic, Billings, Montana, United States

IPD SHARING:
Plan to Share IPD: No